CLINICAL TRIAL: NCT00619554
Title: Zogenix Intraject Instructions for Use Pilot Study
Brief Title: A Study on the Intraject Instructions for Use
Status: Completed | Type: Observational
Sponsor: Zogenix, Inc. (Industry)
Responsible Party: Steve Farr, PhD., Zogenix, Inc.
Organization: UCB Pharma (Industry)
Other Study IDs: ZX000-0702
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2008-02

CONDITIONS: Healthy
Keywords: Healthy volunteers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is designed to create an instruction set simple enough to be understood by migraine subjects as they were experiencing miagraine attacks.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Written Informed Consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers from the community
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2007-07; Primary Completion 2007-08 (Actual)